CLINICAL TRIAL: NCT00408252
Title: A Phase II Study Of Su011248 In Patients With Recurrent And/Or Metastatic Squamous Head And Neck Carcinoma.
Brief Title: Efficacy of SU 011248 in Head And Neck Carcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Too frequent grade 3-4 toxicities
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2006-01; IIR Study A6181004
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Recurrent Disease; Squamous Cell Head and Neck Carcinoma; Palliative Treatment
Keywords: recurrent or locally advanced; cytokine failure
MeSH Terms: conditions — Recurrence; Squamous Cell Carcinoma of Head and Neck | interventions — Biopsy; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): patients will receive SU011248 in monotherapy
  Interventions: Other: biopsies; Drug: SU011248

INTERVENTIONS:
Other: biopsies — No intervention, only biopsy for translational project
Drug: SU011248 — no intervention

SUMMARY:
Preclinical studies as well as phase I and II trials have demonstrated that SU11248 has antitumor activity in renal cell carcinoma, breast cancer, neuroendocrine tumor and GIST. So at the light of these pre-clinical and clinical data, it seems interesting and promising to test SU011248 in these poor prognosis patients.

DETAILED DESCRIPTION:
This is an open-label phase II, multicenter study. Eligible patients will receive SU011248 in monotherapy (37.5 mg given continuously without interruption). Tumor check-up will be performed every 6-8 weeks. Treatment will be continued until disease progression or unacceptable toxicities according to the patient or the investigator (the median for treatment in renal cell study was 8 months).

Since, head and neck tumors are easily accessible for iterative biopsy, this study will offer the opportunity to get tumor biopsies before and after SU011248. Our study will allow translational research with biopsies at crucial timing: at baseline before any treatment, , during the treatment with SU011248 (cycle 1, between week 4 and 6), for patients with stable disease or partial response, a new biopsy will be performed at the time of disease progression to try to understand the mechanisms of tumor or resistance.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent and/or metastatic head and neck squamous cell carcinoma not amenable to curative treatment with surgery and/or chemotherapy and/or radiation
* Recurrence must be confirmed by anatomopathology (cytology or biopsy)
* At least one measurable lesion by MRI or CT-scan
* Failed or relapsing after first line chemotherapy including a platinum* or a taxane-based chemotherapy regimen
* Patients ineligible for chemotherapy could be included in first line
* ECOG performance status 0 -2, in stable medical condition
* Patients must be able to swallow tablets
* Patients must have an expected survival of at least 3 months
* Paraffin-embedded tumor tissue available for immunohistochemistry
* Patients must be over 18 years old and must be able to give written informed consent
* Women of child-bearing age must have a negative pregnancy test
* Female patients of child-bearing age must use effective contraception until 3 months have elapsed after the last injection
* Patients must have normal organ function
* For patients with local recurrence and easily accessible tumors, acceptance of iterative biopsies to store tumor samples (Formaldehyde for immunochemistry, RNA later)
* Acceptance of giving 20 ml of blood for eventual pharmacogenomic analysis
* Acceptance of giving two plasma samples (3ml) at baseline and after 4 weeks of treatment with SU011248
* Signed informed consent prior to beginning protocol specific procedure

Exclusion Criteria:

* Non-squamous head and neck cancer
* Nasopharynx cancer
* Brain metastases
* More than two lines of chemotherapy for palliative treatment (except if chemotherapy was given as a part of a multimodal treatment given with a curative intent)
* Surgery or irradiation or investigational drugs within 4 weeks before study inclusion
* Other uncontrolled illnesses (active infections requiring antibiotics, bleeding disorders, …)
* Active uncontrolled coronary disease or cardiac insufficiency (Ejection fraction below 40%)
* Previous malignancy, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Other concomitant anticancer therapies
* Previous treatment with anti-VEGF, PDGF, or kit therapies. EGFR therapy is not an exclusion criteria.
* Organic brain syndrome or significant psychiatric abnormality that would preclude participation in the full protocol and follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-02; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of SU011248 alone in patients with head and neck cancer in term of overall response rate (RECIST, see statistical consideration) | every 6 weeks

SECONDARY OUTCOMES:
Determine the safety profile of SU011248 alone in patients with head and neck cancer. | untill disaese progression
Determine the efficacy of SU011248 alone in patients with head and neck cancer: progression-free survival and survival. | untill disease progression
Translational research objective:To better understand the mechanisms of sunitinib resistance by the analysis of the tumor biopsies (RNA, gene expression profile) and protein profile (plasma samples). Exploratory analyses. | at week 6 and at disaese progression after recist response

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pascal H Machiels, MD PhD, Principal Investigator — Cliniques Universitaires St Luc
Locations (9):
- Belgium (3):
  - Cliniques Universiatires St LUC UCL, Brussels
  - clinique Sainte Elisabeth, Namur
  - Clinique universiataire de Mont Godinnes UCL, Yvoir
- France (6):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre G-f Leclerc, Dijon
  - Centre Alexis Vautrin, Nancy
  - René Gauducheau, Saint-Herblain
  - CHU Bretonneau, Tours
  - Institut Gustave Roussy, Villejuif